CLINICAL TRIAL: NCT06200818
Title: Clinical, Radiographic and Patient's Acceptance
Brief Title: Clinical, Radiographic and Patient Acceptance Evaluation of LASER Compared to Formocresol Pulpotomies inPrimary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Hamdy, Lecturer of pediatric dentistry and dental public health, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecD061519
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Pulpitis Reversible
Keywords: Pulp, vital pulp therapy, pulpotomy, formocresol, diode, erbium
MeSH Terms: interventions — Lasers, Semiconductor; formocresol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Formocresol (Active Comparator)
  Interventions: Procedure: Formocresol
- Diode laser (Experimental)
  Interventions: Procedure: Diode laser
- Er:CrYSGG (Experimental)
  Interventions: Procedure: Er:CrYSGG

INTERVENTIONS:
Procedure: Diode laser
  Arms: Diode laser
Procedure: Er:CrYSGG
  Arms: Er:CrYSGG
Procedure: Formocresol
  Arms: Formocresol

SUMMARY:
The goal of this clinical trial was to compare the clinical and radiographic success of laser versus formocresol pulpotomy in primary molars. The main questions it aimed to answer was:

• Does laser pulpotomy has higher clinical and radiographic success rate as formocresol pulpotomy in primary molars?

Participants were selected according to eligibility criteria to undergo pulpotomy for their lower primary molars under local anesthesia using one of the following techniques:

* Group 1: Formocresol
* Group 2: Diode laser Group 3: Er:CrYSGG laser Clinical and radiographic follow up were performed for 18 months

DETAILED DESCRIPTION:
In all teeth, local anaesthesia was administered using 7.0 mg/kg 4% articane + 1: 100,000 epinephrine (with a maximum total dosage of 500 mg)

- Rubber dam isolation was done.

Access cavity preparation:

* In all groups, caries removal was done with a sterile #330 high-speed bur, and coronal access cavity preparation was done with a sterile #4 high-speed round bur using high speed hand piece and water coolant. The access cavity was then refined using a sterile high-speed fissure bur. LASER operating parameters: Figure (10)

  * Wavelength: 2780 nm
  * Repetition rate: 15 Hz
  * Water spray: 80
  * Air : 60
  * Emission mode: Free-running pulsed
  * Tip: MZ 10- 6 mm, Zip Tip
  * Average power: 8 Watt The coronal pulp was amputated by a sterile sharp excavator, the amputated sites were rinsed with water. Hemorrhage was controlled by placing sterile, saline- wetted cotton pellets on the radicular pulp stumps under slight pressure (Thompson et al., 2001) for 5 min for primary hemostasis ( J Dent Res 84(12) 2005). At this stage, the achievement of complete hemostasis was an inclusion criterion. If bleeding recommenced afterwards, partial pulpectomy was performed and the tooth was excluded from the study.
* After achieving complete haemostasis pulp stumps were treated according to each group: Group1: (control group)
* A cotton pellet that was moistened with 1:5 diluted bottle of FC (Formacresol, PREVEST DenPro, Digiana, Jammu, India) was placed over the pulp stumps for 5 minutes. After removal of the cotton, the fixed pulp stumps were capped with reinforced zinc oxide and eugenol base (Zinconol, PREVEST DenPro, Digiana, Jammu, India). Group2: (Diode LASER group)
* All patients, parents and clinical staff were requested to wear appropriate eye protection goggles during laser application, Figure (12). After achieving hemostasis, pulp stumps was treated with Diode LASER (980 nm).If hemostasis was not achieved, the process was repeated one more time until adequate hemostasis was achieved, Figure (15, 16). Diode LASER radiation (wavelength 980 nm) was delivered to the canal orifices with a special handpiece and fiber glass of 200 μm diameter, Figure (13), the parameters were set at: Figure (14) Emission mode: Pulsed contact mode Time: 2 seconds. Power: 2 Watt power with average power of 1 Watt and total energy of one spot, corresponding to two minutes and 31 seconds exposure was 4.0 J/cm 2. Group3: (Erbium:Chromium,YSGG LASER group) Pulp tissues in this group were treated with Erbium:Chromium,YSGG LASER (2780 nμ). (Waterlase Biolase®, Biolase, Inc., San Clemente, California, USA) Once the pulp chamber was opened, the laser tip was placed into the pulp chamber using for approximately 15 seconds. In most instances, this was repeated three times. If hemostasis was not achieved, the process was repeated one more time until adequate hemostasis was achieved. Er: Cr, YSGG LASER radiation (wavelength 2780 nμ) was delivered with a special handpiece, and a tip: MZ 10- 6 mm, Zip Tip, to the canal orifices.

LASER operating parameters:

* Wavelength: 2780 nm
* Repetition rate: 50 Hz
* Water spray: 1
* Air : 20
* Emission mode: Free-running pulsed In all groups, reinforced zinc oxide eugenol cement was placed over the pulp stumps, and the tooth was restored with a stainless steel crown. Preoperative and postoperative as well as follow up periapical radiographs at 6, 12 and18 months were obtained by standardized paralleling technique and exposure time of 0.25 seconds. An XCP film holder (Super Bite, Hawe Neos DentalSA, Switzerland) was used. Digital radiographs were obtained and scanned using size 0 phosphostimulable phosphor plates [X mind AC (de Gotzen, Italy) and Fona-Scaneo, phosphor plate scanner, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical criteria One or more primary teeth indicated for pulpotomy due to carious pulp exposure. No spontaneous pain No swelling No tenderness to percussion No pathological mobility No sinus tract opening No initially unsuccessful hemorrhage control. 2. Radiographic criteria Teeth without inter-radicular radiolucency No loss of lamina dura or widened periodontal ligament space No physiologic root resorption of more than one-third.

Exclusion Criteria:

* Clinical mobility Spontaneous pain Swelling Tenderness to percussion Pathological mobility Non restorable teeth. Teeth with necrotic pulp. Pre-operative radiographic pathology such as resorption, periradicular or furcal radiolucency, a widened periodontal ligament space, or physiological root resorption of more than one-third. Parents / Patients not willing to be a part of the study. Any kind of medical history contraindicating the pulp treatment.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-12-20 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical and radiographic success | 18 months
  Clinical success criteria:
  1. Restoration intact;
  2. No pain or tenderness;
  3. No mobility;
  4. No swelling;
  5. No fistula;
  6. No gingival inflammation-represented by pain, redness, or bleeding-around the tooth/crown. Radiographic success at follow-up visits should meet the following criteria:
  1. No external root resorption; 2. No internal root resorption; 3. No inter-radicular bone resorption. 4. No Widening of the periodontal ligament space. 5. No periapical bone resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Hamdy, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No